CLINICAL TRIAL: NCT01955551
Title: A Randomized Controlled Trial Evaluating the Use of Motivational Interviewing to Increase Engagement by Low-income Parents in Preventive Parenting-skills Programming
Brief Title: Motivational Interviewing to Increase Parent Engagement in Preventive Parenting Programming
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Julie Lumeng, Associate Professor of Pediatrics, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SDBP_Research_Grant_2013
Record Dates: First submitted 2013-09-28; First posted 2013-10-07 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Behavior Problems; Parent-Child Relations
MeSH Terms: conditions — Mental Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motiv. Interviewing (Experimental): In the MI (motivational interviewing) study arm, participants will receive MI phone calls designed to evoke change talk and to prompt the participant to identify goals in regards to child behavior or parenting. The caller will engage in problem solving with the participants.
  Interventions: Behavioral: Motivational Interviewing
- Anticipatory Guidance (Active Comparator): In the Anticipatory Guidance on Child Development study arm, the participants will receive two phone calls with no MI content. The content of these phone calls is derived from an alignment of the Teaching Strategies GOLD® standards with the Head Start Development and Early Learning Framework. , This content is entirely scripted and pre-specified.
  Interventions: Behavioral: Anticipatory Guidance on Child Development

INTERVENTIONS:
Behavioral: Motivational Interviewing — In the Motivational Interviewing study arm, participants will receive MI phone calls designed to evoke change talk and to prompt the participant to identify goals in regards to child behavior or parenting. The caller will engage in problem solving with the participants.
  Arms: Motiv. Interviewing
Behavioral: Anticipatory Guidance on Child Development — In the Anticipatory Guidance on Child Development study arm, the participants will receive two phone calls with no MI content. The content of these phone calls is derived from an alignment of the Teaching Strategies GOLD® standards with the Head Start Development and Early Learning Framework. , This content is entirely scripted and pre-specified.
  Arms: Anticipatory Guidance

SUMMARY:
Evidence-based programs aimed at enhancing parenting skills are effective, and pediatricians identify many parents who could benefit from such programs. Low-income children have high rates of behavior problems and their family system and environmental exposures often lead to cumulative and daunting levels of risk for poor functional outcomes; their parents are highly likely to benefit from parenting supports. However, low-income families are the most likely to drop out of parenting interventions, meaning the families and children with the greatest need receive the least support. Fewer than 25% of low-income families recruited to parenting programs will participate in even one session, and only about half of these parents will participate in more than half of the sessions offered. The aims of this trial are:

Aim 1: To test the hypothesis that the provision of motivational interviewing (MI), as compared to an attention control (AC) condition, will increase the engagement of low-income parents of preschoolers in an evidence-based parenting skills group (the Incredible Years Series (IYS)). For this study, the outcome of engagement is operationally defined as intention to attend IYS sessions, attendance, and satisfaction with the IYS program.

Aim 2: To test the hypothesis that the effect of MI on engagement in IYS will be impacted by the following moderators: parenting self-efficacy, child behavior problems, and maternal depression.

The investigators hypothesize that the effect of MI on engagement will be greater among parents with lower parenting self-efficacy and parents of children with more behavior problems, but less among parents with more maternal depressive symptoms.

The investigators will use a stratified, randomized controlled trial (RCT) design to evaluate the impact of MI on parent engagement in a well-validated preventive parenting skills intervention, the Incredible Years Series (IYS).

ELIGIBILITY:
Inclusion Criteria:

* all children enrolled in the Head Start agencies involved in this study, who were randomized to the study arm involving the Incredible Years Series

Exclusion Criteria:

* child is a foster child
* parent or child cannot communicate in English

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Participant intention to attend IYS sessions | 1 week

SECONDARY OUTCOMES:
Attendance at initial IYS session | 1 month
Number of IYS sessions attended | 9 months
Satisfaction with the IYS program, as measured by a 46-item IYS questionnaire | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Julie C Lumeng, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States